CLINICAL TRIAL: NCT05806437
Title: Patient Blood Management in the Approach to Prosthetic Surgery in Orthopedic
Brief Title: Patient Blood Management in the Approach to Prosthetic Surgery [PBM(L4178)]
Acronym: PBM(L4178)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PBM(L4178)
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-03

CONDITIONS: Anemia, Iron Deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Long assumption (Experimental): Assumpion of SideremilVita for 30 days
  Interventions: Dietary Supplement: sideremil vita cp
- Standard assumption (Active Comparator): Assumpion of SideremilVita for 15 days
  Interventions: Dietary Supplement: sideremil vita cp

INTERVENTIONS:
Dietary Supplement: sideremil vita cp — assunzione per 30 giorni dell'integratore

SUMMARY:
We have been well guided in the "Good use of blood" during major surgery for many years, reaching a percentage of 4% of patients transfused after elective prosthetic operations. Valid patient blood management must provide for the possibility of limiting/zeroing the transfusion risk dependent on preoperative anemia, and the national guideline on PBM (Patient blood management) also underlines this Hypothesis and relevance

DETAILED DESCRIPTION:
We want to analyse patients from a diagnostic point of view (occult blood, diverticulitis, gastrorrhagia) and from the point of view of laboratory parameters (blood count, serum iron, transferrinemia, ferritinemia, transferrin saturation) in ordr to be able to suggest the best approach in preparation to the intervention.

We want to evaluate the effectiveness of this approach, considering the proposed treatments (ferric carboxymaltose, chelated iron, folic acid, sideremil vita) and the transfusion result (or not) obtained

ELIGIBILITY:
Inclusion Criteria:

* Candidates for prosthetic surgery
* Patients of both sexes over 40 years of age
* Hemoglobin values <12 g% for females and 13 g% for males
* % transferrin saturation < 10%
* Willingness and ability to provide informed consent.

Exclusion Criteria:

* Patients with Mediterranean anemia
* Patients with coagulation disorders
* Patients who do not sign the consent form
* Pregnant or breastfeeding women (self-declaration)
* Minor aged

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Reduction in transfusion patients | 7 days post-surgery
  Evaluate the reduction of transfusions in anemic patients treated with SideremilVita for 30 days before the intervention (group B experimental), compared to patients assuming SideremilVita at 15 days before surgery (control group A)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi-Istituto Clinico San Siro, Milan, Italy